CLINICAL TRIAL: NCT05051696
Title: Intra-tumor Injection of Oncolytic Viruses H101 Combined With or Without Radiotherapy in Refractory/Recurrent Gynecological Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Zi (Other)
Responsible Party: Sponsor-Investigator, Liu Zi, Professor, Xi'an Jiaotong University
Organization: Xi'an Jiaotong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LZi
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Genital Neoplasms, Female
Keywords: Cervical Cancer; Ovary Cancer; Endometrial Cancer; Vaginal Neoplasms; Vulvar Neoplasms; H101
MeSH Terms: conditions — Genital Neoplasms, Female; Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncorine (H101) with or without radiotherapy (Experimental): The tumor mass was injected with H101 per day for 5 consecutive days, 3 weeks as one treatment cycle, and 1 to 4 cycles according to the condition of the patient, and the patient was treated with or without radiotherapy in sequential. The injection dose of H101 was determined by the tumor volume or maximum tumor diameter:5.0×10^11 virus particles(VP) for if tumor diameter≤5cm; 1×10^12 VP for the tumor diameter between 5cm and 10cm, and 1.5×10^12 VP for the tumor diameter>10cm.
  Interventions: Drug: H101

INTERVENTIONS:
Drug: H101 — Intra-tumor injected oncolytic viruses H101 within 5 consecutive days,3 weeks for a cycle (1-4cycles)
  Other Names: Radiotherapy

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and safety of oncolytic viruses H101 intra-tumor injection combined with or without radiotherapy in refractory or recurrent gynecological malignancies. And further research the mechanism of oncolytic viruses H101.

DETAILED DESCRIPTION:
Patients with recurrent, radiation/chemotherapy-resistant gynecological cancer carry a poor prognosis. H101 is a recombinant human type-5 adenovirus (Ad5), in which the E1B and E3 gene have been deleted. Previous studies have shown that H101 has anticancer activity and safety in some solid tumors, but has little report in gynecological oncology. In this clinical trial, 60 recurrent or refractory gynecological cancer patients will be enrolled. Based on individual conditions, all eligible patients are intra-tumor injected oncolytic viruses H101 within 5 consecutive days combined with or without radiotherapy in sequential, three weeks for a cycle (1-4 cycles totally). Simultaneously, the tumor sample, peripheral blood, and urine specimen were collected on day1 and day5. Local control rate and side effects are recorded respectively.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at the time of study entry.
* Histological or Cytologically diagnosed gynecological malignancies.
* Failure to prior standard treatment (surgery, chemotherapy, radiotherapy);
* Refractory/recurrence/metastasis gynecological cancer
* At least one measurable lesion according to the RECIST1.1.
* Cooperative Oncology Group-Status (ECOG Status) 0-3.
* The last treatment should be over 2 weeks.

Exclusion Criteria:

* History or evidence of active autoimmune disease that requires systemic treatment.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Patients who have a contraindication to similar drugs.
* That failure to follow up regularly.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Local Control (LC) | 3 months
  LC will be measured from the start date of injection until the date of progressive disease

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year after injection
  ORR is the percentage of participants with presence of complete response (CR), partial response (PR). ORR assessment will be based on RECIST 1.1 criteria
Progress free survival (PFS) | 12 months
  Progress free survival is defined as the time from first day of injection until the first date of either objective disease progression or death due to any cause
adverse events | At day 3, 7 and 30
  Toxicity were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zi Liu, M.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No